CLINICAL TRIAL: NCT01996566
Title: Fatty Acid Taste Thresholds: Caproic, Lauric, Oleic, Linoleic, Linolenic
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Other Study IDs: 055-036
Record Dates: First submitted 2013-08-12; First posted 2013-11-27 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Taste Sensitivity; Fatty Acid Type
Keywords: taste; non-esterified fatty acids; threshold; sensitivity; human
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva will be collected to obtain DNA for analysis of genes for fatty acid receptors and their potential correlation with sensitivity.
Oversight: Data Monitoring Committee: No

SUMMARY:
Differences in human oral sensitivity for caproic, lauric, oleic, linoleic, and linolenic acids will be explored. Prior work indicates that there may be a learning effect in measuring detection thresholds for free fatty acids. This study is designed to determine the number of visits necessary to attenuate this learning effect and also to test whether this effect continues across different types of fatty acids or is specific to each fatty acid. This will aid in understanding how many visits are required to obtain reliable data and if less expensive fatty acids can be used to attenuate learning before testing thresholds for more expensive fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* in good health
* available for 3 months

Exclusion Criteria:

* Participation in a different fat taste study in previous 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals between 18 and 60 years of age from any ethnic background who are in good health and are available for the next three months will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Oral sensitivity to oleic, lauric, linoleic, linolenic and caproic acids measured by the ascending 3 alternative forced choice test as described in American Society and Testing and Methods E679 | Measured at weekly intervals over 3 months
  Thresholds for taste of each fatty acid will be determined using the 3 alternative forced choice test. Participants will taste 3 samples, one of which contains a fatty acid, and select which sample they believe is different. The concentration of fatty acid used will range from very dilute to a maximum of 5%. The test is repeated over the range of concentrations until a participant is able to correctly identify the fatty acid or until the maximum concentration is reached.

SECONDARY OUTCOMES:
DNA sequence of potential fatty acid receptors (e.g., CD36, GPR120, GPR48) | This will be collected at the final visit of the study, approximate 2-3 months from participant enrollment depending on how frequently the participant is able to come to the lab
  Saliva will be collected to analyze any correlations between fatty acid receptor genes and sensitivity.
Amount of habitual dietary fat intake | Baseline
  A survey will be administered to determine each participant's habitual dietary fat intake
Measurement of hunger | This will be measured at every study visit (21 visits plus 1 screening visit) over the 2-3 months of the study
  Participants will rate how hungry they are on a line scale because commencing each study threshold test

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Running CA, Mattes RD. Different oral sensitivities to and sensations of short-, medium-, and long-chain fatty acids in humans. Am J Physiol Gastrointest Liver Physiol. 2014 Aug 1;307(3):G381-9. doi: 10.1152/ajpgi.00181.2014. Epub 2014 Jun 12. PMID 24924750